CLINICAL TRIAL: NCT00543049
Title: Phase II Trial in Platinum-refractory Ovarian Cancer: A Randomized Multicenter Trial With SU11248 to Evaluate Dosage, Tolerability, Toxicity and Effectiveness of a Multitargeted Receptor Tyrosine Kinase Inhibitor Monotherapy
Brief Title: Randomized Multicenter Trial With SU11248 Evaluating Dosage,Tolerability,Toxicity and Effectiveness of a Multitargeted Receptor Tyrosine Kinase Inhibitor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AGO Study Group (Other)
Collaborators: Philipps University Marburg (Other); HSK Reasearch GmbH Wiesbaden (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGO-OVAR 2.11
Record Dates: First submitted 2007-10-10; First posted 2007-10-12 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Platinum Refractory Epithelial Ovarian Cancer; Primary Cancer of the Peritoneum; Cancer of the Fallopian Tube
Keywords: platinum refractory; epithelial ovarian cancer; primary cancer of the peritoneum; cancer of the fallopian tube
MeSH Terms: conditions — Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 non-continuous (Other): Subjects will receive open-label sunitinib = SU11248 at a dose of 50.0 mg once daily. After 28 days, treatment will be paused for 14 days and cycle one is completed, followed by resumption of therapy as cycle one for up to one year (therapy can be continued in case of tumor response and benefit for the patient for more than one year).
  Interventions: Drug: Sunitinib
- 2 continuous (Other): Subjects will receive open-label sunitinib = SU11248 at a dose of 37.5 mg once daily continuously. Treatment period up to one year (therapy can be continued in case of tumor response and benefit for the patient for more than one year).
  Interventions: Drug: SUNITINIB

INTERVENTIONS:
Drug: Sunitinib — Sunitinib, oral, 50mg once daily, 28 days then paused for 14 days, for up to one year
  Other Names: Sutent, Sunitinib, SU011248
  Arms: 1 non-continuous
Drug: SUNITINIB — Sunitinib, oral, 37,5 mg once daily continuously, up to one year
  Other Names: SUTENT, Sunitinib, SU011248
  Arms: 2 continuous

SUMMARY:
Ovarian cancer is most often recognized in advanced clinical state, the initial therapeutic strategies consist of a platinum containing chemotherapy subsequent to primary surgery. Although initially responsive to platinum-paclitaxel containing chemotherapy, a significant number of patients will show tumor progression during first line chemotherapy or relapse within six months after completion of first line chemotherapy, therefore being characterized as chemotherapy resistant. Any second line chemotherapy will result in approximately 10% of overall response, underlining the poor prognosis for these patients with an estimated median overall survival of 20 weeks.

In addition to conventional chemotherapeutics, so called small molecules are of high interest to establish new strategies in chemotherapy-refractory ovarian cancer (and in the long run first line chemotherapy). SU11248 is a polytargeting tyrosine kinase inhibitor.

SU11248 has demonstrated clinical efficacy in kidney cancer and GIST, further clinical trials have been initiated in other tumor entities. Growth pattern and biological targets present in ovarian cancer indicate that SU11248 might be a promising compound for the treatment of ovarian cancer. Especially, VEGFR, PDGFR and c-kit are specific targets for SU11248, which are expressed in ovarian cancer. The different targets of SU11248 provide a potential advantage of this compound compared to single-target molecules in chemotherapy-refractory ovarian cancer.

DETAILED DESCRIPTION:
This study in patients with ovarian cancer refractory to platinum based chemotherapy is designed as a randomized, 2-schedule and dose-level, open-label, multicenter phase II study to select the better dose and schedule arm for further investigation.

72 patients will be randomized in a 1:1 ratio to receive oral SU11248 therapy either 37.5 mg/day continuously or 50mg/day for 4 weeks followed by 14 days off.

Patients will get outpatients treatment. At screening the patients' eligibility will be assessed, their baseline and demographic characteristics obtained, and the baseline values for the effect variables collected. Patients with measurable lesions as well as non-measurable disease will be included into this trial. Measurable lesion will be documented by CT or MRI scan and CA-125 values, non-measurable lesions will be monitored by analysis of CA°125 levels.

The patients' safety will be monitored during and up to 30 days after termination of SU11248 therapy.

In patients with measurable lesions at baseline, the (post)-treatment values for effect according to the RECIST criteria will be collected as shown in table 6. In case of CR or PR, a confirmatory CT or MRI scan is required after an interval of at least four weeks. Antitumor effects according to CA°125 levels will be determined in the same time intervals and, in addition, 28 days after last SU11248 application in patients with CA°125 response according to GCIG guidelines during therapy.

For post study follow-up, patients and/or their physicians will be contacted via phone for overall survival and TTP (including the method of diagnosis and additional treatment) every 2 months for their life time.

ELIGIBILITY:
Inclusion Criteria:

* Women, 18 years and older, written (signed and dated) informed consent
* Histological confirmed epithelial ovarian cancer, primary cancer of the peritoneum or fallopian tube
* Up to three prior chemotherapies, at least one platinum based chemotherapy
* Platinum refractory or resistant ovarian cancer (defined as stable (SD) or progressive disease (PD) during platinum containing chemotherapy, or treatment free interval < 6 months after stop of platinum based chemotherapy)
* Measurable or non-measurable disease
* Elevated CA°125 level (> 2 x ULN in case of normal CA°125 after prior chemotherapy; or ≥ 2 x nadir CA°125 value after prior chemotherapy, when CA° 125 levels remained elevated above normal) in case of non-measurable disease
* ECOG performance status 0-2
* Negative pregnancy test within 5 days before randomization and adequate contraception in women with childbearing potential

Adequate organ function as defined by the following criteria:

* Serum aspartate aminotransferase (AST; serum glutamate-oxalate transferase [SGOT]) and serum alanine aminotransferase (ALT; serum glutamate-pyruvate transferase [SGPT]) <=2.5 x upper limit of normal (ULN). If liver function abnormalities are due to underlying malignancy, then AST and ALT may be <=5x ULN
* Total serum bilirubin <=1.5 x ULN
* Prothrombin time (PT) and partial thromboplastin time (PTT) <=1.5 x ULN
* Serum albumin >= 3.0 g/dL
* Absolute neutrophil count (ANC) >=1500/µl
* Platelets >=100,000/µl
* Hemoglobin >=9.0 g/dL
* Serum creatinine <=1.5 x ULN
* TSH within normal range Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures Resolution of all toxic effects of any prior chemotherapy, surgical procedures, radiotherapy, or other cancer related therapies to NCI CTCAE (Version 3.0) grade >=1 and to the baseline laboratory values as defined in inclusion criterion (see before)

Exclusion Criteria:

* Borderline tumor of the ovaries
* Acute or chronic infection
* Any required concurrent cancer chemotherapy or antineoplastic endocrine therapy or radiotherapy
* Exposure to investigational trial medication, cancer chemo- or radiotherapy within the last 28 days prior to start of study treatment
* Known or suspected hypersensitivity to investigational compound
* Second malignancy interfering with prognosis of the patient
* Cachectic patients with a body weight <45 kg
* Patients requiring parenteral nutrition
* Patients with ileus within the last 28 days
* Any of the following within the 12 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, pulmonary embolism, deep vein thrombosis, or other thromboembolic event
* Current treatment with therapeutic doses of anticoagulant
* Current treatment with CYP3A4 inhibitors or -inducers
* Hypertension that cannot be controlled by medications (>150/100 mmHg despite optimal medical therapy)
* Ongoing cardiac dysrhythmias of NCI CTCAE grade >=2, atrial fibrillation of any grade, or prolongation of the QTc interval to >470 msec for females

  * Left ventricular ejection fraction (LVEF) <=50% as measured by echocardiogram
  * NCI CTCAE Grade 3 hemorrhage within 4 weeks of starting study treatment
* Evidence of neurological signs/symptoms suggestive of brain metastases, spinal cord compression, or new evidence of brain or leptomeningeal disease
* Known human immunodeficiency virus (HIV) positivity or acquired immunodeficiency syndrome (AIDS)-related illness
* Patients with any other severe concurrent disease, which is an undue risk for the patient by participating in the present study
* Any further condition which according to the investigator results in an undue risk of the patient by participating in the present study
* Major surgery, radiation therapy, or systemic therapy within 3 weeks of first study treatment. At least 7 days should elapse from the time of minor surgical procedure including placement of an access device or fine needle aspiration before randomization into this study can occur.
* Wounds that have not completely healed, active ulcer(s), or bone fracture(s).
* Prior high-dose chemotherapy requiring hematopoietic stem cell rescue.
* Prior radiation therapy to >25% of the bone marrow.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2007-09; Primary Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
objective response rate | one year

SECONDARY OUTCOMES:
tolerability and toxicity, overall survival, duration of response, time to progression, stable disease | one year

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Wagner, MD, PhD, Principal Investigator — Universitätsklinikum Gießen u. Marburg, Klinik f. Gynäkologie, Gyn. Endokrinologie u. Onkologie
Locations (16):
- Germany (16):
  - Malterser-Krankenhaus Bonn-Rhein/Sieg, Frauenklinik, Bonn
  - Klinikum Bremen-Mitte gGmbH, Frauenklinik, Bremen
  - Universitätsklinikum Carl Gustav Carus, Klinik u. Poliklinik für Frauenheilkunde und Geburtshilfe, Dresden
  - Universitätsklinikum, Universitätsfrauenklinik, Essen
  - Klinikum der JWG Universität Frankfurt, Universitätsfrauenklinik, Frankfurt am Main
  - Universitätsklinikum Freiburg, Department Universitäts-Frauenklinik, Freiburg im Breisgau
  - Klinikum der Ernst-Moritz-Universität, Klinik u. Poliklinik für Gyn. - u. Geb.Hilfe, Greifswald
  - Med. Hochschule Hannover, Frauenklinik, Hanover
  - St. Vincentius Kliniken AG, Frauenklinik, Karlsruhe
  - Universitätsklinikum Schleswig-Holstein Campus Kiel, Klinik f. Gynäkologie u. Geburtshilfe, Kiel
  - Otto-von-Guericke-Universität, Klinik für Frauenheilkunde und Geburtshilfe, Magdeburg
  - Universitätsklinikum Gießen u. Marburg, Standort Marburg, Klinik f. Gynäkologie, Gyn. Endokrinologie u. Onkologie, Marburg
  - Elblandkliniken Meißen-Radebeul GmbH, Gynäkologie, Radebeul
  - Universitätsklinikum Tübingen, Frauenklinik, Tübingen
  - Universitätsklinikum, Universitätsfrauenklinik, Ulm
  - Dr. Horst Schmidt Kliniken GmbH, Klinik f. Gynäkologie u. Gyn. Onkologie, Wiesbaden

REFERENCES:
- [Result] Baumann KH, du Bois A, Meier W, Rau J, Wimberger P, Sehouli J, Kurzeder C, Hilpert F, Hasenburg A, Canzler U, Hanker LC, Hillemanns P, Richter B, Wollschlaeger K, Dewitz T, Bauerschlag D, Wagner U. A phase II trial (AGO 2.11) in platinum-resistant ovarian cancer: a randomized multicenter trial with sunitinib (SU11248) to evaluate dosage, schedule, tolerability, toxicity and effectiveness of a multitargeted receptor tyrosine kinase inhibitor monotherapy. Ann Oncol. 2012 Sep;23(9):2265-2271. doi: 10.1093/annonc/mds003. Epub 2012 Feb 29. PMID 22377563
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961